CLINICAL TRIAL: NCT07179952
Title: A Study to Evaluate Efficacy and Safety of Slow Release DHEA
Brief Title: Efficacy and Safety of Slow Release Dehydroepiandrosterone (DHEA )
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kirsten Kloepfer, Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26427; P01HL158507 (NIH)
Record Dates: First submitted 2025-08-06; First posted 2025-09-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Intervention Model Description: placebo controlled crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy will maintain mask
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Slow Release DHEA (Active Comparator): Subjects will take active capsule 1/day for 4 weeks
  Interventions: Drug: Slow Release DHEA
- Placebo (Placebo Comparator): Subjects will take placebo capsule 1/day for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Slow Release DHEA — Slow-release dehydroepiandrosterone capsule
  Other Names: dehydroepiandrosterone
  Arms: Slow Release DHEA
Drug: Placebo — placebo capsule
  Arms: Placebo

SUMMARY:
There is evidence to suggest that DHEA-based treatment could be beneficial to patients with asthma, yet one of the main treatments for asthma (taking glucocorticoids, a hormone that is effective in reducing inflammation), suppresses the production of DHEA.

In this study, the investigators want to test and evaluate the safety of DHEA-based treatment.

DETAILED DESCRIPTION:
During this study, participants will come to the study site 4-5 times and have 2 telephone visits over a period of approximately 3 months. Participants will complete the following:

Informed Consent: Coordinators will explain the study to participants. If participants decide to participate, they will be asked to review, sign, and date the consent form.

Medical History: Coordinators will review participants medical chart and record relevant medical history, including the history of asthma, other pertinent respiratory details, and any information regarding underlying diseases such as cystic fibrosis or chronic lung disease. Coordinators will also ask participants about any medications they are currently taking.

Demographic Information: Coordinators will collect information about participants such as age, gender, and race.

Physical Exam & Vital Signs: The study doctor will examine the participants head, eyes, ears, nose, throat; heart, chest, lungs, and abdomen; extremities and skin; and any other areas as appropriate for any abnormal signs and symptoms. In addition, they will also check participants vital signs which includes measuring blood pressure, temperature, heart rate, breathing rate, pulse oximetry (the amount of oxygen in the blood), and height and weight.

Urine Samples: All participants will be asked to provide a urine sample that will be tested for cotinine levels (to indicate whether participant has been exposed to nicotine recently).

Pregnancy Testing & Contraception Females who can get pregnant will also have a pregnancy test. Because DHEA is a hormone and it is not known how it will affect a developing baby, if the participant is pregnant, they cannot be in this study. Additionally, they must practice a medically acceptable form of contraception during study participation. Medically acceptable contraceptives include: (1) surgical sterilization, (2) approved hormonal contraceptives such as birth control pills, (3) barrier methods (such as a condom or diaphragm) used with a spermicide, (4) abstinence, or (5) an intrauterine device (IUD).

Blood Samples: At each in-person visit, the study team will draw up to 40ml (about 8 teaspoons) of the participants blood to assess overall blood health (complete blood count, or CBC), metabolic and organ function (comprehensive metabolic panel), hormone levels, and immune system activity (cytokine responses and peripheral blood mononuclear cells or PBMCs). The study team will also use the participants blood sample for genotyping (studying genetic makeup), their ability to process DHEA; and measuring the level of DHEA-S. For male subjects, a portion will be used for a Prostate Specific Antigen Test, which checks for prostate cancer.

Spirometry: This test measures how much air a persons lungs can hold and how fast they can breathe out. Participants will take a deep breath and then blow into a mouthpiece as hard as possible and for as long as possible. They might have to wear soft nose clips during the test to stop air from escaping through the nose. They will be asked to repeat this test at least 3 times. They will be asked to take a bronchodilator (a medication that relaxes and opens the airways in the lungs) such as albuterol while completing spirometry during some study visits. The study team will provide the bronchodilator used for the test.

Methacholine Challenge Testing (MCT): This test will be done only if the participant failed to demonstrate 10% reversibility in Forced Expiratory Volume in 1 Second (FEV1) and there are no historical MCT results available.

MCT is done to confirm that the participant has asthma. Methacholine is approved by the FDA. When methacholine is inhaled, it causes the airways to spasm (contract involuntarily) and narrow if asthma is present. During this test, the participant will inhale increasing amounts of methacholine aerosol mist before and after spirometry. The MCT is considered positive, meaning asthma is present, if the participants lung function drops by at least 20%.

If the participants airways tighten at any point, they will be given albuterol to open their airways. Often, the staff person doing the test will know that the participants airways are tightening before they feel it, by seeing a drop in the test results. A bronchodilator is always given at the end of the test to reverse the effects of the methacholine.

Completion of Questionnaire & Symptom Diary: Participants will be asked to complete the Asthma Control Test (ACT) and the Asthma Control Questionnaire (ACQ) at several study visits. They will also be asked to complete a medication dosing and symptom diary at home between visits 1 and 3 and visits 4 and 6.

Randomization: Participants will be randomly assigned (like flipping a coin) to receive either DHEA or placebo.

Study Drug: DHEA is an over-the-counter supplement that is available on the market without prescription. In this study, the participants will be taking DHEA or placebo as a capsule that has been formulated in a specific way that the investigators expect will make it as effective as possible. The participants will be provided enough capsules for the four-week window of administration.

At Visits 3 and 6, the participants will please return all unused DHEA capsules and packaging to the study team.

There is also one unscheduled visit that will be used in case the participant needs to return to the study site for any reason to finish study activities.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female age ≥ 18 and ≤ 50 years at the time of enrollment
2. Evidence of asthma demonstrated by reversibility at visit 0 or by historical methacholine or bronchodilator reversibility if testing was performed under either the 2017 European Respiratory Society (ERS) technical standard (22) or the 1999 American Thoracis Society (ATS) Guidelines (23) or outside studies, provided that full sets of flow volume loops have been reviewed and approved by the PI. These criteria are defined as one of the following:

   1. For bronchodilator reversibility: An increase in FEV1 ≥ 10% (24) compared to the baseline (and 200 ml) after up to 8 puffs of albuterol
   2. For historical methacholine responsiveness: Positive methacholine defined as Provocative Concentration of Methacholine causing a 20% fall in FEV1 (PC20) ≤ 16 mg/ml, or Provocative Dose of Methacholine causing a 20% fall in FEV1 (PD20) ≤ 400 mcg
3. Physician diagnosis of asthma according to NHLBI guidelines
4. Consistent use of an Inhaled Corticosteroids (ICS) inhaler for the prior 2 months
5. Non-smoker
6. Females must not be pregnant or breastfeeding
7. Absence of non-allergic comorbidities

Exclusion Criteria:

1. Pregnant or actively trying to become pregnant; breastfeeding
2. Positive urine pregnancy test
3. Known lung disease other than asthma
4. Acute (non-asthma related) dyspnea, viral respiratory illness or asthma exacerbation within 4 weeks of screening
5. Systemic glucocorticoid dosing for maintenance >10 mg/day of prednisone or equivalent
6. Patients with significant non-allergic comorbidities (e.g. cerebral palsy, heart disease, kidney disease, liver disease, etc.)
7. Patients with any know central or peripheral endocrine abnormality such as precocious puberty or diabetes
8. Patients with any known previous adverse reaction to DHEA
9. Current smoker or pack year history > 5 years (includes vaping/nicotine inhalation devices)
10. Positive urine cotinine test (> 100 mg/mL)
11. Use of prednisone or antibiotics in the last 4 weeks
12. Use of any performance-enhancing drugs in the last 2 weeks
13. Use of DHEA in the last 2 weeks
14. Androgen use for any reason.
15. Any other condition or finding that would compromise the safety of the subject or the quality of the study data, or otherwise interfere with achieving the study objectives, as determined by the PI
16. Menopausal amenorrhea by history
17. Positive Prostate-Specific Antigen (PSA) (>4 ng/ml) test
18. Prior diagnosis of vocal cord dysfunction, bronchopulmonary dysplasia, cystic fibrosis, chronic obstructive pulmonary disorder, or other lung disease
19. Systolic blood pressure > 150 mm Hg and/or diastolic blood pressure >90 mm Hg
20. Heart rates outside the range of 50 to 120 beats per minutes or with a pathologic irregularity
21. Patients afflicted with any additional acute or chronic pathology that in the opinion of the screening physician makes them unsuitable for study or increases the risks associated with the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Scores of Asthma Control Test | From baseline to 12 hours after the final dose of final arm (up to 94 days)
  Determine if slow-release DHEA in patients with asthma improves asthma control based on ACT (Asthma Control Test) scoring. Results will be between 0-25.
  20-25: Well-controlled asthma 16-19: Not well-controlled asthma 15 or less: Very poorly-controlled asthma
Scores of Asthma Control Questionnaire | From baseline to 12 hours after the final dose of final arm (up to 94 days)
  Determine if slow-release DHEA in patients with asthma improves asthma control based on ACQ (Asthma Control Questionnaire) scoring. Results will be between 0 and >1.5.
  Well-controlled asthma is indicated by a score ≤ 0.75 Partly controlled asthma is indicated by a score between 0.75 to < 1.5 Not well-controlled asthma is indicated by a score ≥ 1.5

SECONDARY OUTCOMES:
Measurements of Forced Expiratory Volume in 1 Second | From baseline to 12 hours after the final dose of final arm (up to 94 days)
  FEV1 (Forced Expiratory Volume in 1 Second) will be measured using spirometry at baseline and every in person visit.
Measurements of Fractional Exhaled Nitric Oxide | From baseline to 12 hours after the final dose of final arm (up to 94 days)
  FeNO (Fractional Exhaled Nitric Oxide) will be measured at baseline and at each in person visit.
Incidences of Adverse Events | From baseline to 12 hours after the final dose of final arm (up to 94 days)
  Adverse Events will be recorded from baseline and at every visit.

REFERENCES:
- [Background] Shimizu M, Matsuzawa A, Iwaguchi T. Analysis of splenic lymphocytes with high electrophoretic mobility in adult and aged nude mice. J Immunol Methods. 1985 Nov 28;84(1-2):95-103. doi: 10.1016/0022-1759(85)90418-1. PMID 2866215
- [Background] Ehrenspeck G. Effect of 3-isobutyl-1-methylxanthine on HCO3- transport in turtle bladder. Evidence for electrogenic HCO3- secretion. Biochim Biophys Acta. 1982 Jan 22;684(2):219-27. doi: 10.1016/0005-2736(82)90009-8. PMID 6173069
- [Background] Soffer RL. Peptide acceptors in the arginine transfer reaction. J Biol Chem. 1973 Apr 25;248(8):2918-21. No abstract available. PMID 4572514
- [Background] Arieff AI, Armstrong DK. Parathyroid hormone and uremic neurotoxicity: an unproven association. Contrib Nephrol. 1980;20:56-66. doi: 10.1159/000384954. No abstract available. PMID 6995013
- [Background] Rupp H. Modulation of tension generation at the myofibrillar level -- an analysis of the effect of magnesium adenosine triphosphate, magnesium, pH, sarcomere length and state of phosphorylation. Basic Res Cardiol. 1980 Mar-Apr;75(2):295-317. doi: 10.1007/BF01907579. No abstract available. PMID 6967310
- [Background] Lahm T, Albrecht M, Fisher AJ, Selej M, Patel NG, Brown JA, Justice MJ, Brown MB, Van Demark M, Trulock KM, Dieudonne D, Reddy JG, Presson RG, Petrache I. 17beta-Estradiol attenuates hypoxic pulmonary hypertension via estrogen receptor-mediated effects. Am J Respir Crit Care Med. 2012 May 1;185(9):965-80. doi: 10.1164/rccm.201107-1293OC. Epub 2012 Mar 1. PMID 22383500
- [Background] Warren AP, Pasternak CA. Common pathway for the induction of hexose transport by insulin and stress. J Cell Physiol. 1989 Feb;138(2):323-8. doi: 10.1002/jcp.1041380215. PMID 2645305
- [Background] de Crespigny LC, Robinson HP, Quinn M, Doyle L, Ross A, Cauchi M. Ultrasound-guided fetal blood transfusion for severe rhesus isoimmunization. Obstet Gynecol. 1985 Oct;66(4):529-32. PMID 3931012
- [Background] Hammond GR, Thomas GJ. Failure to reactivate the septal syndrome in rats. Physiol Behav. 1971 May;6(5):599-601. doi: 10.1016/0031-9384(71)90212-5. No abstract available. PMID 5149451
- [Background] Bulitta JB, Jiao Y, Drescher SK, Oliver A, Louie A, Moya B, Tao X, Wittau M, Tsuji BT, Zavascki AP, Shin BS, Drusano GL, Sorgel F, Landersdorfer CB. Four Decades of beta-Lactam Antibiotic Pharmacokinetics in Cystic Fibrosis. Clin Pharmacokinet. 2019 Feb;58(2):143-156. doi: 10.1007/s40262-018-0678-x. PMID 29936678
- [Background] Bailey E. Regulation of hepatic lipid metabolism during development of the rat. Biochem Soc Trans. 1981 Oct;9(5):371-2. doi: 10.1042/bst0090371. No abstract available. PMID 6456955
- [Background] Deal WB. The settling froth. J Fla Med Assoc. 1979 Sep;66(9):910. No abstract available. PMID 479800
- [Background] Hunt JF, Fang K, Malik R, Snyder A, Malhotra N, Platts-Mills TA, Gaston B. Endogenous airway acidification. Implications for asthma pathophysiology. Am J Respir Crit Care Med. 2000 Mar;161(3 Pt 1):694-9. doi: 10.1164/ajrccm.161.3.9911005. PMID 10712309
- [Background] Carraro S, Doherty J, Zaman K, Gainov I, Turner R, Vaughan J, Hunt JF, Marquez J, Gaston B. S-nitrosothiols regulate cell-surface pH buffering by airway epithelial cells during the human immune response to rhinovirus. Am J Physiol Lung Cell Mol Physiol. 2006 May;290(5):L827-32. doi: 10.1152/ajplung.00406.2005. PMID 16603595
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Background] Watson AC, Rosenfield RL, Fang VS. Recovery from glucocorticoid inhibition of the responses to corticotrophin-releasing hormone. Clin Endocrinol (Oxf). 1988 May;28(5):471-7. doi: 10.1111/j.1365-2265.1988.tb03681.x. PMID 2850875
- [Background] Jollin L, Thomasson R, Le Panse B, Baillot A, Vibarel-Rebot N, Lecoq AM, Amiot V, De Ceaurriz J, Collomp K. Saliva DHEA and cortisol responses following short-term corticosteroid intake. Eur J Clin Invest. 2010 Feb;40(2):183-6. doi: 10.1111/j.1365-2362.2009.02219.x. Epub 2009 Oct 29. PMID 19874391
- [Background] Brehm R. [Chronic pyelonephritis, pregnancy and the incidence of pregnancy toxemias]. Wien Klin Wochenschr. 1967 Feb 24;79(8):145-8. No abstract available. German. PMID 5597997
- [Background] Rossmann I, Korber F, Siegmund P. [An apparatus for maintaining the constancy of low substrate concentrations in kinetic measurements with the pH-Stat]. Z Klin Chem Klin Biochem. 1970 May;8(3):269-72. No abstract available. German. PMID 5470749
- [Background] Coates AL, Wanger J, Cockcroft DW, Culver BH; Bronchoprovocation Testing Task Force: Kai-Hakon Carlsen; Diamant Z, Gauvreau G, Hall GL, Hallstrand TS, Horvath I, de Jongh FHC, Joos G, Kaminsky DA, Laube BL, Leuppi JD, Sterk PJ. ERS technical standard on bronchial challenge testing: general considerations and performance of methacholine challenge tests. Eur Respir J. 2017 May 1;49(5):1601526. doi: 10.1183/13993003.01526-2016. Print 2017 May. PMID 28461290
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836
- [Background] Stanojevic S, Kaminsky DA, Miller MR, Thompson B, Aliverti A, Barjaktarevic I, Cooper BG, Culver B, Derom E, Hall GL, Hallstrand TS, Leuppi JD, MacIntyre N, McCormack M, Rosenfeld M, Swenson ER. ERS/ATS technical standard on interpretive strategies for routine lung function tests. Eur Respir J. 2022 Jul 13;60(1):2101499. doi: 10.1183/13993003.01499-2021. Print 2022 Jul. PMID 34949706
- [Background] Prefaut C. [Effects of oral almitrine on gas exchange in chronic respiratory insufficiency and hypercapnia]. Rev Fr Mal Respir. 1980;8(6):587-97. No abstract available. French. PMID 6794117
- [Background] Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med. 1999 Jan;159(1):179-87. doi: 10.1164/ajrccm.159.1.9712108. PMID 9872837
- [Background] Hunt PJ, Gurnell EM, Huppert FA, Richards C, Prevost AT, Wass JA, Herbert J, Chatterjee VK. Improvement in mood and fatigue after dehydroepiandrosterone replacement in Addison's disease in a randomized, double blind trial. J Clin Endocrinol Metab. 2000 Dec;85(12):4650-6. doi: 10.1210/jcem.85.12.7022. PMID 11134123
- [Background] Brooke AM, Kalingag LA, Miraki-Moud F, Camacho-Hubner C, Maher KT, Walker DM, Hinson JP, Monson JP. Dehydroepiandrosterone improves psychological well-being in male and female hypopituitary patients on maintenance growth hormone replacement. J Clin Endocrinol Metab. 2006 Oct;91(10):3773-9. doi: 10.1210/jc.2006-0316. Epub 2006 Jul 18. PMID 16849414
- [Background] Binder G, Weber S, Ehrismann M, Zaiser N, Meisner C, Ranke MB, Maier L, Wudy SA, Hartmann MF, Heinrich U, Bettendorf M, Doerr HG, Pfaeffle RW, Keller E; South German Working Group for Pediatric Endocrinology. Effects of dehydroepiandrosterone therapy on pubic hair growth and psychological well-being in adolescent girls and young women with central adrenal insufficiency: a double-blind, randomized, placebo-controlled phase III trial. J Clin Endocrinol Metab. 2009 Apr;94(4):1182-90. doi: 10.1210/jc.2008-1982. Epub 2009 Jan 6. PMID 19126625
- [Background] Sahelian R, Borken S. Dehydroepiandrosterone and cardiac arrhythmia. Ann Intern Med. 1998 Oct 1;129(7):588. doi: 10.7326/0003-4819-129-7-199810010-00020. No abstract available. PMID 9758585
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880

DOCUMENTS (2):
  • Study Protocol (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT07179952/Prot_000.pdf
  • Informed Consent Form (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT07179952/ICF_001.pdf